CLINICAL TRIAL: NCT06055452
Title: Effects and Mechanism of SGLT2 Inhibitors in Pre-heart Failure Populations With Hypertension
Brief Title: Effects of SGLT2 Inhibitors in Pre-heart Failure Populations With Hypertension
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-GSP-GG-18
Record Dates: First submitted 2023-09-14; First posted 2023-09-26 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pre-Heart Failure; Hypertension
Keywords: Pre-Heart Failure; Hypertension; Randomized controlled trial; Empagliflozin
MeSH Terms: conditions — Hypertension | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Each participant in the empagliflozin treatment group takes a daily dose of 10mg.
  Other Names: Jardiance®
  Arms: Empagliflozin
Drug: Placebo — Each participant in the placebo group takes matching placebo.
  Arms: Placebo

SUMMARY:
In this multicenter, randomized, placebo-controlled trial in pre-heat failure patients with hypertension and without diabetes, we will enroll 120 eligible patients to randomized to receive placebo or engagliflozin (10mg/d) for follow them for 6 months. The primary endpoint is the left atrial volume index, which reflects left ventricular diastolic function. We sought to comprehensively evaluate the effect of engagliflozin on the structure and function and explore its underlying mechanisms.

DETAILED DESCRIPTION:
Hypertension is the leading risk factor of heart failure with preserved heart failure. The overall control rate is about 16% in China. Given the large amounts of hypertensive patients at pre-heart failure (stage B), it's critical to explore the effect of additional cardioprotective medication in addition to well-controlled blood pressure. Sodium-glucose cotransporter-2 inhibitors (engagliflozin) have been shown to improve cardiac function or prognosis in patients with diabetes or heart failure. However, whether it has a cardioprotective effect on hypertensive patients with pre-heart failure and without diabetes remains unknown. We will conduct a multicenter, randomized, placebo-controlled trial in pre-heat failure patients with hypertension and without diabetes. We will enroll 120 eligible patients randomized to receive a placebo or engagliflozin (10mg/d) for follow them for 6 months. The primary endpoint is the left atrial volume index, which reflects left ventricular diastolic function. The secondary endpoints include echocardiography or magnetic resonance imaging to measure structural and functional parameters, blood pressure, glucose, and blood biomarkers of inflammation and fibrosis. We sought to comprehensively evaluate the effect of empagliflozin on the structure and function and explore the underlying mechanisms to provide insights and evidence for the prevention of heart failure in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

• Meeting all the following criteria:

1. Aged 40 and above; less than 75 years.
2. Hypertensive patients currently taking at least one antihypertensive medication as recommended by guidelines, and blood pressure is within the target range (<140/90 mmHg).
3. The left atrial volume index measured by transthoracic echocardiography exceeds 34 mL/m², or the ratio of the average E/e' >9 and left atrial volume index >= 29 mL/m² measured by transthoracic echocardiography.
4. Signing an informed consent form.

Exclusion Criteria:

* • Exclusion criteria include any of the following conditions:

  1. History of diabetes.
  2. History of heart failure.
  3. History of coronary artery disease.
  4. Left ventricular systolic dysfunction, defined as LVEF < 50%.
  5. Systolic blood pressure < 100 mmHg.
  6. A history of arrhythmias such as atrial fibrillation, atrial flutter, frequent atrial premature contractions, and frequent ventricular premature contractions may impact the structural and functional aspects of the heart.
  7. Moderate and above valvular heart disease.
  8. Severe obstructive disease of the left ventricular outflow tract, including aortic valve stenosis.
  9. Visited within the past 1 month due to Genitourinary tract infection.
  10. Chronic kidney disease or estimated Glomerular Filtration Rate (eGFR) < 45 ml/min/1.73m².
  11. Alanine aminotransferase or aspartate aminotransferase levels > 3 times the upper limit of normal.
  12. Contraindications to taking SGLT2 inhibitors.
  13. Currently taking SGLT2 inhibitors, SGLT-1/2 inhibitors, or other antihyperglycemic medications (including metformin, glucagon-like peptide-1 receptor agonists, etc.).
  14. Pregnancy or planning pregnant, or currently breastfeeding.
  15. Malignant tumors or other severe illnesses with a life expectancy of less than 3 years.
  16. History of alcohol abuse or substance abuse within the past year.
  17. Mental disorders or communication barriers, cognitive impairments, or other severe illnesses that may affect participation in the study.
  18. Participation in or currently participating in other clinical trials within the last 3 months.
  19. Known poor compliance with study follow-up or study drug.
  20. Any condition or contraindication that makes a person intolerant to magnetic resonance imaging (MRI) or contraindicates MRI examination, such as the presence of implanted intracranial aneurysm clips, cardiac pacemakers or defibrillators, insulin pumps, etc.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of left atrial volume index | 6 months
  Changes in Left Atrial Volume Index (LAVI, mL/m2) as measured by MRI from baseline to 6 months.

SECONDARY OUTCOMES:
Change of cardiac structure and functional | 6 months
  1. Left ventricular functional indicators: Echocardiography/Magnetic Resonance Imaging measured Left Ventricular Ejection Fraction (LVEF, %), the ratio of early mitral inflow velocity to early diastolic mitral annular velocity (E/e', cm/s), and Global Longitudinal Strain (GLS, %).
  2. Left ventricular structural indicators: Echocardiography/Magnetic Resonance Imaging measured Left Ventricular Mass Index (LVMI, g/m2).
  3. Left atrial functional indicators: Echocardiography/Magnetic Resonance Imaging measured Left Atrial Ejection Fraction (LAEF, %) and echocardiography measured Left Atrial Volume Index (LAVI, mL/m2).
Biomarkers | 6 months
  Biomarker concentrations were measured as follows:
  1. NT-pro BNP in picograms per milliliter (pg/mL).
  2. Cardiac Troponin I in nanograms per milliliter (ng/mL).
  3. Cardiac Fibrosis Biomarkers, including Collagen type I alpha 1 (Col1A1) in nanograms per milliliter, Matrix Metalloproteinases (MMP-2, MMP-3, MMP-4) in picograms per milliliter (pg/mL) and soluble ST2 protein (sST-2) in nanograms per milliliter (ng/mL).
  4. Inflammation Biomarkers, including High-sensitivity C-reactive protein (hs-CRP) in milligrams per liter (mg/L) and Interleukin-6 (IL-6), Interleukin-1β (IL-1β), and Galectin-3 (Gal-3) in picograms per milliliter (pg/mL).
Estimated Glomerular Filtration Rate (eGFR) | 6 months
  Change of eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zheng, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (2):
- China (2):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medial Sciences, Shenzhen, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No